CLINICAL TRIAL: NCT00529516
Title: Observer Blind Study to Evaluate Safety, Reactogenicity and Immunogenicity of GSK Biologicals Influenza Vaccine GSK576389A Administered to Adults Over 65 Years Previously Vaccinated With the Same Vaccine, Compared to Fluarix™
Brief Title: Evaluate Safety & Immunogenicity of GSK Bio's Influenza Vaccine GSK576389A After Repeated Vaccination in Elderly Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109821
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Results first posted 2012-05-30 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Fluarix; GSK Bio's influenza vaccine GSK576389A; Influenza infection
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- FluAS25 Group (Experimental): Subjects aged 65 years and above, who had received one dose of GlaxoSmithKline (GSK) Biologicals' AS25 adjuvanted influenza vaccine (GSK576389A) in study NCT00377585, received one dose of GlaxoSmithKline (GSK) Biologicals' AS25 adjuvanted influenza vaccine (GSK576389A) in the current study.
  Interventions: Biological: GSK Biologicals Influenza Vaccine GSK576389A
- Fluarix ≥ 65 years age Group (Active Comparator): Subjects aged 65 years and above, who had received one dose of Fluarix™ vaccine in study NCT00377585, received one dose of Fluarix™ vaccine in the current study.
  Interventions: Biological: Fluarix
- Fluarix 18-40 years age Group (Active Comparator): Subjects aged between 18 and 40 years, who had received one dose of Fluarix™ vaccine in study NCT00377585, received one dose of Fluarix™ vaccine in the current study.
  Interventions: Biological: Fluarix

INTERVENTIONS:
Biological: Fluarix — Single dose, Intramuscular injection
  Arms: Fluarix 18-40 years age Group; Fluarix ≥ 65 years age Group
Biological: GSK Biologicals Influenza Vaccine GSK576389A — Single dose, Intramuscular injection
  Arms: FluAS25 Group

SUMMARY:
Since influenza vaccines are administered every year because of the frequent change in their antigenic composition, the safety and immunogenicity profile of GSK Biologicals' influenza vaccine GSK576389A will be re-evaluated after repeated vaccine administration. In this observer blind study, the subjects previously enrolled in study 104888 (NCT00377585) will receive a dose with the 2007-2008 season's formulations of Fluarix or GSK576389A. Only subjects who were previously enrolled in study 104888 (NCT00377585) are eligible for participation in this study.

DETAILED DESCRIPTION:
This study involves 2 age groups (based on primary study):

Subjects enrolled in the >= 65 yrs age group in the primary study. Subjects enrolled in the 18-40 yrs age group in the primary study. The study will be conducted in an open manner for this age group.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical evaluation before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.
* Male or female subjects who participated in the 104888 study (NCT00377585) and were enrolled in the >= 65 years age group or in the 18-40 years age group .

Exclusion Criteria:

* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study.
* Planned administration of a vaccine not foreseen by the study protocol up to 30 days after vaccination
* Planned administration of an influenza vaccine other than the study vaccines during the entire study period
* Any vaccination against influenza since January 2007
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of hypersensitivity to a previous dose of influenza vaccine
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s)
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or pre-existing laboratory screening tests
* Acute disease at the time of enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to vaccination, or planned use during the study period
* Any medical conditions in which IM injections are contraindicated
* Pregnant or lactating female, or planning to become pregnant or to discontinue contraceptive precautions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1252 (Actual)
Dates: Start 2007-10-15; Primary Completion 2007-12-21 (Actual); Study Completion 2008-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (9):
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
- GSK Investigational Site, Ghent, Belgium
- Germany (8):
  - GSK Investigational Site, Messkirch, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Langquaid, Bavaria
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
- Norway (7):
  - GSK Investigational Site, Bekkestua
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Fredrikstad
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Haugesund
  - GSK Investigational Site, Skien

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 109821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109821 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Started | 475 | 488 | 289
Completed | 472 | 486 | 288
Not Completed | 3 | 2 | 1
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group | Total
Number analyzed (Participants) | 475 | 488 | 289 | 1252
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.8 (5.50) | 73.7 (5.80) | 30.9 (6.64) | 63.86 (19.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 253 | 167 | 668
  Male | 227 | 235 | 122 | 584

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Solicited local AEs assessed include ecchymosis, pain, redness and swelling. Any: any symptom regardless of intensity grade. Grade 3 pain: considerable pain at rest, which prevented normal everyday activities. Grade 3 ecchymosis, redness and swelling: more than 100 millimeter.
Time Frame: During a 7-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort on subjects who completed the symptom sheet.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 472 | 487 | 288
Subjects
  Any Ecchymosis | 7 | 7 | 2
  Grade 3 Ecchymosis | 0 | 0 | 0
  Any Pain | 271 | 76 | 170
  Grade 3 Pain | 2 | 0 | 0
  Any Redness | 111 | 14 | 16
  Grade 3 Redness | 12 | 0 | 0
  Any Swelling | 44 | 8 | 7
  Grade 3 Swelling | 1 | 0 | 0

2. Primary Outcome: Duration of Solicited Local Adverse Events
Description: Duration was expressed as the median number of days the symptom was experienced.
Time Frame: During a 7-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, on subjects that reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 271 | 76 | 170
Days
  Ecchymosis (N= 7; 7; 2) | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 5.0] | 4.5 [4.0 to 5.0]
  Pain (N= 271; 76; 170) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 5.0]
  Redness (N= 111; 14; 16) | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 1.5 [1.0 to 3.0]
  Swelling (N= 44; 8; 5) | 3.0 [1.0 to 7.0] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Adverse Events (AEs)
Description: Solicited general AEs assessed include arthralgia, fatigue, headache, myalgia, nausea, shivering and fever. Any: any symptom regardless of intensity grade; any fever: oral temperature greater than or equal to 38 degrees Celsius (°C). Grade 3: symptoms that prevented normal activity ; Grade 3 fever: oral temperature greater than 40°C. Related: symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 7-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort on subjects who completed the symptom sheet.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 472 | 487 | 288
Subjects
  Any Arthralgia | 80 | 34 | 23
  Grade 3 Arthralgia | 2 | 0 | 1
  Related Arthralgia | 65 | 20 | 22
  Any Fatigue | 131 | 46 | 71
  Grade 3 Fatigue | 4 | 0 | 1
  Related Fatigue | 109 | 29 | 54
  Any Headache | 102 | 49 | 54
  Grade 3 Headache | 4 | 1 | 1
  Related Headache | 87 | 37 | 39
  Any Myalgia | 132 | 51 | 70
  Grade 3 Myalgia | 4 | 0 | 1
  Related Myalgia | 116 | 38 | 64
  Any Nausea | 35 | 23 | 17
  Grade 3 Nausea | 2 | 0 | 0
  Related Nausea | 29 | 15 | 13
  Any Shivering | 95 | 31 | 31
  Grade 3 Shivering | 5 | 0 | 0
  Related Shivering | 88 | 24 | 28
  Any Fever | 17 | 0 | 1
  Grade 3 Fever | 0 | 0 | 0
  Related Fever | 15 | 0 | 1

4. Primary Outcome: Duration of Solicited General Adverse Events
Description: Duration was expressed as the median number of days the symptom was experienced.
Time Frame: During a 7-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, on subjects that experienced the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 132 | 51 | 70
Days
  Arthralgia (N= 80; 34; 23) | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Fatigue (N= 131; 46; 71) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Headache (N= 102; 49; 54) | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Myalgia (N= 132; 51; 70) | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 6.0]
  Nausea (N= 35; 23; 17) | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 4.0]
  Shivering (N= 95; 31; 31) | 1.0 [1.0 to 5.0] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 6.0]
  Fever (N= 17; 0; 1) | 1.0 [1.0 to 2.0] | NA [NA to NA] — No Fever was experienced by any of the subjects in this arm. | 1.0 [1.0 to 1.0]

5. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any: any AE regardless of intensity or relationship to vaccination. Grade 3: AE that prevented normal activity. Related: AE considered by the investigator to be causally related to the study vaccination.
Time Frame: During a 21-day follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort which included all subjects with study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 475 | 488 | 289
Subjects
  Any AEs | 82 | 68 | 62
  Grade 3 AEs | 7 | 5 | 5
  Related AEs | 19 | 6 | 11

6. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the vaccination phase of the study (Day 0 to Day 20) and during the long term follow-up phase of the study (Day 21 to Day 179)
Population: The analysis was performed on the Total Vaccinated Cohort which included all subjects with study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 475 | 488 | 289
Subjects
  Any SAEs - Vaccination Phase | 2 | 3 | 1
  Related SAEs - Vaccination Phase | 1 | 0 | 0
  Any SAEs - Long Term Follow-up Phase | 21 | 24 | 3
  Related SAEs - Long Term Follow-up Phase | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Any and Related Medically Significant Conditions (MSCs)
Description: Medically significant conditions assessed include conditions prompting emergency room visits, hospitalizations or physician visits.
Time Frame: as for outcome 6
Population: The analysis was performed on the Total Vaccinated Cohort which included all subjects with study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 475 | 488 | 289
Subjects
  Any MSCs - Vaccination Phase | 22 | 25 | 11
  Grade 3 MSCs - Vaccination Phase | 3 | 3 | 2
  Related MSCs - Vaccination Phase | 1 | 1 | 1
  Any MSCs - Long Term Follow-up Phase | 112 | 137 | 71
  Grade 3 MSCs - Long Term Follow-up Phase | 23 | 29 | 20
  Related MSCs - Long Term Follow-up Phase | 0 | 0 | 1

8. Secondary Outcome: Serum Hemagglutination-inhibition (HI) Antibody Titers Against Each of the Three Vaccine Strains
Description: Titers were expressed as Geometric Mean Titers. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the According-to-Protocol (ATP) Cohort for immunogenicity haemagglutination-inhibition (HI) which included all evaluable subjects who complied with the protocol up to the end of the active phase, for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 447 | 461 | 271
Titer
  A/Solomon Islands [Day 0] (N= 445; 461; 270) | 10.5 [9.6 to 11.5] | 10.8 [9.9 to 11.9] | 48.9 [39.9 to 59.9]
  A/Solomon Islands [Day 21] (N= 447; 461; 271) | 103.5 [92.4 to 115.8] | 53.7 [47.6 to 60.7] | 143.4 [125.8 to 163.6]
  A/Wisconsin [Day 0] (N= 445; 461; 270) | 110.0 [97.7 to 123.9] | 79.5 [70.5 to 89.7] | 112.5 [98.1 to 129.0]
  A/Wisconsin [Day 21] (N= 447; 461; 271) | 430.6 [394.0 to 470.6] | 217.9 [196.3 to 241.8] | 251.2 [226.4 to 278.8]
  B/Malaysia [Day 0] (N= 445; 461; 270) | 95.8 [86.8 to 105.7] | 82.5 [75.2 to 90.6] | 110.5 [95.9 to 127.2]
  B/Malaysia [Day 21] (N= 447; 461; 271) | 202.2 [187.1 to 218.5] | 152.3 [140.0 to 165.6] | 209.2 [188.9 to 231.7]

9. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against Each of the Three Vaccine Strains
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below1:10 and a post-vaccination titer greater than or equal to1:40 or a pre-vaccination titer greater than or equal to1:10 and at least a four-fold increase in post-vaccination titer. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: At Day 21
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 445 | 461 | 270
Subjects
  A/Solomon Islands | 320 | 238 | 94
  A/Wisconsin | 226 | 156 | 66
  B/Malaysia | 82 | 66 | 46

10. Secondary Outcome: Seroconversion Factors for HI Antibodies Against Each of the Three Vaccine Strains
Description: Seroconversion factor was defined as the fold increase in serum HI Geometric Mean Titers post-vaccination compared to Day 0.
Time Frame: At Day 21
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 445 | 461 | 270
Fold increase
  A/Solomon Islands | 9.8 [8.7 to 11.1] | 5.0 [4.4 to 5.5] | 2.9 [2.5 to 3.4]
  A/Wisconsin | 3.9 [3.5 to 4.3] | 2.7 [2.5 to 3.0] | 2.2 [2.0 to 2.5]
  B/Malaysia | 2.1 [2.0 to 2.3] | 1.8 [1.7 to 2.0] | 1.9 [1.7 to 2.1]

11. Secondary Outcome: Number of Subjects Seroprotected for HI Antibodies Against Each of the Three Vaccine Strains
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to1:40 that is usually accepted as indicating protection. The three vaccine strains assessed included A/Solomon Islands, A/Wisconsin and B/Malaysia.
Time Frame: At Days 0 and 21
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 447 | 461 | 271
Subjects
  A/Solomon Islands [Day 0] (N= 445; 461; 270) | 71 | 73 | 164
  A/Solomon Islands [Day 21] (N= 447; 461; 271) | 381 | 306 | 255
  A/Wisconsin [Day 0] (N= 445; 461; 270) | 381 | 362 | 235
  A/Wisconsin [Day 21] (N= 447; 461; 271) | 445 | 442 | 270
  B/Malaysia [Day 0] (N= 445; 461; 270) | 392 | 399 | 236
  B/Malaysia [Day 21] (N= 447; 461; 271) | 445 | 443 | 268

12. Secondary Outcome: Number of Cluster of Differentiation 4 (CD4) T-cells (Per Million CD4 T-cells) Producing at Least 2 Different Immune Markers
Description: Results are presented as the geometric mean number of immune response marker-positive CD4 T-cells (per million CD4 T-cells) for pooled vaccine strains. Immune markers assessed include Cluster of Differentiation 40 Ligand (CD40L), interleukin-2 (IL-2), tumor necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ).
Time Frame: At Day 0 and 21
Population: The analysis was performed on the ATP cohort of immunogenicity Cell-Mediated Immunity (CMI) which included a subset of subjects from the ATP Cohort for immunogenicity HI. This included subjects for whom data for immune response marker-positive CD4 result was available 21 days after vaccination.
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 65 | 63 | 40
Cells per million
  Day 0 (N= 62; 60; 39) | 830.72 (889.90) | 674.91 (567.07) | 1276.25 (701.42)
  Day 21 (N= 65; 63; 40) | 2013.28 (1388.55) | 1010.22 (1069.96) | 1607.66 (839.45)

13. Secondary Outcome: Number of CD4 T-cells (Per Million CD4 T-cells) Producing at Least CD40L and Another Immune Marker
Description: Results are presented as the geometric mean number of CD40L-positive CD4 T-cells (per million CD4 T-cells) for pooled vaccine strains. Other immune markers assessed include interleukin-2 (IL-2), tumor necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ).
Time Frame: At Day 0 and 21
Population: as for outcome 12
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 65 | 63 | 40
Cells per million
  Day 0 (N= 62; 60; 39) | 822.37 (875.39) | 660.01 (560.95) | 1260.65 (681.46)
  Day 21 (N= 65; 63; 40) | 1961.18 (1337.11) | 981.82 (1056.18) | 1556.00 (830.54)

14. Secondary Outcome: Number of CD4 T-cells (Per Million CD4 T-cells) Producing at Least IFN-γ and Another Immune Marker
Description: Results are presented as the geometric mean number of IFN-γ -positive CD4 T-cells (per million CD4 T-cells) for pooled vaccine strains. Other immune markers assessed include Cluster of Differentiation 40 Ligand (CD40L), interleukin-2 (IL-2) and tumor necrosis factor alpha (TNF-α).
Time Frame: At Day 0 and 21
Population: as for outcome 12
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 65 | 63 | 40
Cells per million
  Day 0 (N= 62; 60; 39) | 513.25 (586.78) | 371.64 (397.45) | 753.45 (556.25)
  Day 21 (N= 65; 63; 40) | 1081.11 (966.36) | 574.28 (685.03) | 870.84 (589.37)

15. Secondary Outcome: Number of CD4 T-cells (Per Million CD4 T-cells) Producing at Least IL-2 and Another Immune Marker
Description: Results are presented as the geometric mean number of IFN-γ -positive CD4 T-cells (per million CD4 T-cells) for pooled vaccine strains. Other immune markers assessed include Cluster of Differentiation 40 Ligand (CD40L), tumor necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ).
Time Frame: At Day 0 and 21
Population: as for outcome 12
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 65 | 63 | 40
Cells per million
  Day 0 (N= 62; 60; 39) | 769.96 (809.58) | 634.57 (518.17) | 1030.23 (585.91)
  Day 21 (N= 65; 63; 40) | 1644.34 (1110.14) | 856.60 (855.82) | 1288.54 (664.82)

16. Secondary Outcome: Number of CD4 T-cells (Per Million CD4 T-cells) Producing at Least TNF-α and Another Immune Marker
Description: Results are presented as the geometric mean number of IFN-γ -positive CD4 T-cells (per million CD4 T-cells) for pooled vaccine strains. Other immune markers assessed include Cluster of Differentiation 40 Ligand (CD40L) and interferon gamma (IFN-γ).
Time Frame: At Day 0 and 21
Population: as for outcome 12
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 65 | 63 | 40
Cells per million
  Day 0 (N= 62; 60; 39) | 586.39 (698.83) | 409.05 (415.62) | 746.02 (551.82)
  Day 21 (N= 65; 63; 40) | 1189.34 (945.05) | 608.51 (700.32) | 921.15 (549.61)

17. Secondary Outcome: Number of Cluster of Differentiation 8 (CD8) T-cells (Per Million CD8 T-cells) Expressing at Least 2 Different Immune Markers
Description: Results are presented as the geometric mean number of immune response marker-positive CD8 T-cells (per million CD8 T-cells) for pooled vaccine strains. Immune markers assessed include Cluster of Differentiation 40 Ligand (CD40L), interleukin-2 (IL-2), tumor necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ).
Time Frame: At Day 0 and 21
Population: The analysis was performed on the ATP cohort of immunogenicity Cell-Mediated Immunity (CMI) which included a subset of subjects from the ATP Cohort for immunogenicity HI. This included subjects for whom data for immune response marker-positive CD8 result was available 21 days after vaccination.
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 64 | 62 | 40
Cells per million
  Day 0 (N= 55; 54; 39) | 8.25 (166.35) | 6.82 (123.10) | 3.56 (247.08)
  Day 21 (N= 64; 62; 40) | 16.75 (168.54) | 6.51 (112.42) | 3.48 (79.78)

18. Secondary Outcome: Number of CD8 T-cells (Per Million CD8 T-cells) Producing at Least CD40L and Another Immune Marker
Description: Results are presented as the geometric mean number of CD40L-positive CD8 T-cells (per million CD8 T-cells) for pooled vaccine strains. Other immune markers assessed include interleukin-2 (IL-2), tumor necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ).
Time Frame: At Day 0 and 21
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 64 | 62 | 40
Cells per million
  Day 0 (N= 55; 54; 39) | 6.19 (120.88) | 4.33 (134.18) | 2.12 (220.32)
  Day 21 (N= 64; 62; 40) | 8.09 (123.89) | 5.79 (85.20) | 3.64 (71.55)

19. Secondary Outcome: Number of CD8 T-cells (Per Million CD8 T-cells) Producing at Least IFN-γ and Another Immune Marker
Description: Results are presented as the geometric mean number of IFN-γ -positive CD8 T-cells (per million CD8 T-cells) for pooled vaccine strains. Other immune markers assessed include Cluster of Differentiation 40 Ligand (CD40L), interleukin-2 (IL-2) and tumor necrosis factor alpha (TNF-α).
Time Frame: At Day 0 and 21
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 64 | 62 | 40
Cells per million
  Day 0 (N= 55; 54; 39) | 2.77 (69.92) | 2.64 (50.62) | 1.58 (32.08)
  Day 21 (N= 64; 62; 40) | 3.09 (97.36) | 2.82 (56.06) | 2.17 (28.97)

20. Secondary Outcome: Number of CD8 T-cells (Per Million CD8 T-cells) Producing at Least IL-2 and Another Immune Marker
Description: Results are presented as the geometric mean number of IFN-γ -positive CD8 T-cells (per million CD8 T-cells) for pooled vaccine strains. Other immune markers assessed include Cluster of Differentiation 40 Ligand (CD40L), tumor necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ).
Time Frame: At Day 0 and 21
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 64 | 62 | 40
Cells per million
  Day 0 (N= 55; 54; 39) | 6.82 (135.79) | 8.43 (119.70) | 3.21 (249.46)
  Day 21 (N= 64; 62; 40) | 12.70 (159.08) | 5.64 (101.15) | 3.20 (55.75)

21. Secondary Outcome: Number of CD8 T-cells (Per Million CD8 T-cells) Producing at Least TNF-α and Another Immune Marker
Description: Results are presented as the geometric mean number of IFN-γ -positive CD8 T-cells (per million CD8 T-cells) for pooled vaccine strains. Other immune markers assessed include Cluster of Differentiation 40 Ligand (CD40L) and interferon gamma (IFN-γ).
Time Frame: At Day 0 and 21
Population: as for outcome 17
Measure: Geometric Mean (Standard Deviation); unit: Cells per million
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Number analyzed (Participants) | 64 | 62 | 40
Cells per million
  Day 0 (N= 55; 54; 39) | 3.05 (72.38) | 2.48 (42.55) | 3.13 (44.03)
  Day 21 (N= 64; 62; 40) | 5.67 (89.23) | 3.54 (69.71) | 2.73 (40.30)

ADVERSE EVENTS:
Time Frame: Events collected by systematic assessment: 7-day follow-up period after vaccination. Events collected by non-systematic method are reported during the active phase (Day 0 - 20) and during the long term follow-up phase (Day 21 - 179) of the study.
Description: Events collected by systematic assessment are reported for subjects with a symptom diary card available. Events collected by non-systematic method are reported for the Total Vaccinated Cohort.
Arm/Group | FluAS25 Group | Fluarix ≥ 65 Years Age Group | Fluarix 18-40 Years Age Group
Serious Adverse Events (participants affected / at risk) | 23/475 | 27/488 | 4/289
Other Adverse Events (participants affected / at risk) | 346/475 | 162/488 | 200/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FluAS25 Group (N=475) | Fluarix ≥ 65 Years Age Group (N=488) | Fluarix 18-40 Years Age Group (N=289)
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Reported during the active phase of the study (Day 0 - 20)
Chest pain (General disorders) | 0 | 1 | 0 — Reported during the active phase of the study (Day 0 - 20)
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 — Reported during the active phase of the study (Day 0 - 20)
Injection site pain (General disorders) | 1 | 0 | 0 — Reported during the active phase of the study (Day 0 - 20)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — Reported during the active phase of the study (Day 0 - 20)
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Reported during the active phase of the study (Day 0 - 20)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Precursor b-lymphoblastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
Spinal fusion surgery (Surgical and medical procedures) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FluAS25 Group (N=475) | Fluarix ≥ 65 Years Age Group (N=488) | Fluarix 18-40 Years Age Group (N=289)
Pain at the injection site (General disorders) | 271 | 76 | 170
Redness at the injection site (General disorders) | 111 | 14 | 16
Swelling at the injection site (General disorders) | 44 | 8 | 7
Arthralgia (General disorders) | 80 | 34 | 23
Fatigue (General disorders) | 131 | 46 | 71
Headache (General disorders) | 102 | 49 | 54
Myalgia (General disorders) | 132 | 51 | 70
Nausea (General disorders) | 35 | 23 | 17
Shivering (General disorders) | 95 | 31 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.